CLINICAL TRIAL: NCT00762632
Title: An Open-label Phase I/II (Proof of Concept) Trial of an Combination of Nilotinib (AMN 107) and RAD001 in Patients With Acute Myeloid Leukemia
Brief Title: Combination of Nilotinib (AMN107) and RAD001 in Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Prof. Dr. Justus Duyster, Medical faculty of the Technical University Munich
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107ADE01
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: patients with c-kit+ AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — nilotinib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: NILOTINIB — 400 mg Nilotinib bid (total daily dose 800 mg) should be continued 25 weeks
Drug: EVEROLIMUS — Everolimus at 2,5 mg/day should be continued 25 weeks.

SUMMARY:
This is a nonrandomized, open-label study to evaluate the efficacy and safety of combination treatment of Nilotinib and RAD001 in the treatment of c-kit + AML. Patients refractory to standard chemotherapy or not eligible to standard chemotherapy can be included. Patients will be treated with 400 mg Nilotinib bid (total daily dose 800 mg). RAD001 will be added after a treatment duration of 1 week in a dosage of 2,5 mg/day. Treatment duration will be 25 weeks.

ELIGIBILITY:
Inclusion criteria:

1. Patients with:

   * De novo AML or secondary AML from MDS who are not candidates for myelosuppressive chemotherapy, or
   * De novo AML or secondary AML from MDS who have relapsed disease or are refractory to standard therapy
2. Patients at least 18 years or older
3. Patients with WHO performance status of 0 to 2 with a life expectancy under treatment of at least 3 months
4. Patients must have recovered from prior cytotoxic chemotherapy; treatment with Hydroxyurea or Ara-C is allowed until 24 hours to first administration of study drug.
5. Patients must have a serum creatinine of <= 1.5 x ULN, SGOT/SGPT <= 3 x ULN and total bilirubin <= 2.0 x ULN
6. Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
7. Written informed consent obtained according to local guidelines

Exclusion criteria:

1. Patients with AML FAB M3.
2. Patients with an expected doubling of the peripheral blast within one week.
3. Patients who had prior allogeneic, syngeneic, or autologous bone marrow transplant or stem cell transplant less than 2 months previously.
4. Impaired cardiac function, including any one of the following:

   * LVEF < 45% or below the institutional lower limit of the normal range (whichever is higher) as determined by MUGA scan or echocardiogram
   * Complete left bundle branch block
   * Use of a cardiac pacemaker
   * ST depression of > 1mm in 2 or more leads and/or T wave inversions in 2 or more contiguous leads
   * Congenital long QT syndrome dose levels of 400 to 1200 mg QD. Many of the common adverse events reported in the imatinib Phase II leukemia (STI0106, STI0110) studies were also reported in the nilotinib Phase I study, although a notably lower frequency of peripheral edema was identified in the nilotinib study.
   * History of or presence of significant ventricular or atrial tachyarrhythmias
   * Clinically significant resting bradycardia (< 50 beats per minute)
   * QTc > 450 msec on screening ECG (using the QTcF formula)
   * QT prolonging concomitant medication
   * Right bundle branch block plus left anterior hemiblock, bifascicular block
   * Myocardial infarction within 12 months prior to starting Nilotinib
   * Unstable angina diagnosed or treated during the past 12 months
   * Other clinically significant heart disease (e.g., congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
5. Female patients who are pregnant or breast feeding, or adults of childbearing age not employing an effective method of birth control.
6. Concurrent severe and/or uncontrolled medical or psychiatric condition which may interfere with the completion of the study.
7. Patients who had more than 2 prior regimens for their current relapsed or current primary refractory disease
8. Patients with uncontrolled active infection.
9. Patient with any pulmonary infiltrate on the baseline chest X-ray known to be new in the previous 4 weeks. Prior treatment with any investigational drug within the preceding 4 weeks
10. Chronic treatment with systemic steroids or another immunosuppressive agent
11. Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
12. Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
13. Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (i.e., uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, unstable angina, or congestive heart failure - New York Heart Association Class III or IV, ventricular arrhythmias active ischemic heart disease, myocardial infarction within six months, chronic liver or renal disease, active upper GI tract ulceration)
14. A known history of HIV seropositivity
15. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
16. Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except low dose coumarin)
17. Hypokalemia
18. Women who are pregnant or breast feeding, or women able to conceive and unwilling to practice an highly effective method of birth control.
19. Patients who have received prior treatment with an mTor inhibitor.
20. History of noncompliance to medical regimens
21. Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-12; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To determine the rate of hematological response in adult patients with c-kit + AML. state the primary objective of the study | four years

SECONDARY OUTCOMES:
To determine the duration of hematological response. To evaluate overall survival. To evaluate the safety profile of a combination treatment of Nilotinib and RAD001. • To evaluate improvement of symptomatic parameters. • To assess mTor, cKit a | four years

CONTACTS AND LOCATIONS:
Overall Officials: Justus Prof. Duyster, MD, Principal Investigator — Medical faculty of the Technical University Munich
Locations (1):
- Medical faculty of the Technical University Munich, Munich, Bavaria, Germany